CLINICAL TRIAL: NCT00238316
Title: A Randomized Feasibility Study of Letrozole in Postmenopausal Women at Increased Risk for Development of Breast Cancer as Evidenced by High Breast Density
Brief Title: Letrozole in Preventing Breast Cancer in Postmenopausal Women Who Are at Increased Risk for Breast Cancer Due to High Breast Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MAP1; CAN-NCIC-MAP1 (Other: PDQ Identifier); CDR0000445442 (Other: PDQ)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole (Active Comparator)
  Interventions: Drug: letrozole
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: letrozole — 2.5 mg PO daily for 1 year
  Arms: Letrozole
Other: Placebo — 2.5 mg PO daily for one 1 year
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of letrozole may stop cancer from forming or coming back in postmenopausal women who are at increased risk for breast cancer due to high breast density.

PURPOSE: This randomized phase II trial is studying how well letrozole works in preventing breast cancer in postmenopausal women who are at increased risk for breast cancer due to high breast density.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the proportion of postmenopausal women who are at increased risk for the development or recurrence of breast cancer, based on high breast density (≥ grade 4), who achieve a decrease in breast density of ≥ 1 grade after treatment with letrozole for 1 year.

Secondary

* Determine whether a decrease in breast density grade is sustained at 1 year in patients treated with this drug.
* Correlate plasma estrogen profile (E1, E1S, E2) with breast density grade at baseline in these patients.
* Determine the percentage of patients with breast tissue hyperplasia and atypical hyperplasia, as assessed by histopathological examination of breast tissue biopsies, before and after treatment with this drug.
* Determine the changes in estrogen profile from baseline, at 1 year, and 1 year after cessation of this drug in these patients.
* Compare changes in predetermined specific parameters of safety at the end of 1 year of treatment with this drug with baseline evaluations of these patients.
* Determine whether modifications of these predetermined specific parameters of safety are sustained 1 year after cessation of treatment with this drug in these patients.
* Determine the general safety of 1 year of treatment with this drug in these patients.
* Compare the effects of this drug on menopause-specific quality of life of these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to breast density grade (4/6 vs 5/6 vs 6/6). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral letrozole once daily for 1 year in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily for 1 year in the absence of unacceptable toxicity.

Menopause-specific quality of life is assessed at baseline and then at 12 and 24 months.

After completion of study treatment, patients are followed at 6 months and 1 year.

PROJECTED ACCRUAL: A total of 120 patients (80 in arm I and 40 in arm II) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk for the development or recurrence of breast cancer, as defined by 1 of the following:

  * Baseline mammogram indicating mammographic density occupying ≥ 25% (grade 4/6, 5/6, or 6/6) of the breast tissue

    * No suspicion of breast cancer, unless subsequently ruled out
  * Prior ductal carcinoma in situ (DCIS)

    * Untreated disease OR > 6 months since completion of adjuvant endocrine therapy
    * Receptor status of lesion is not required
  * Prior invasive breast cancer

    * Breast cancer must have been surgically removed at time of original diagnosis with no evidence of metastases
* No clinical evidence of breast cancer
* Acceptable quality dual-energy x-ray absorptiometry (DEXA) of the L2-L4 postero-anterior (PA) spine and hip performed within past 6 months

  * Bone mass density T-score of either PA spine or hip must be ≥ 2.0 SD below the mean peak bone mass in young normal woman
* Stable chronic leukemia allowed
* Hormone receptor status:

  * Hormone receptor-negative, -positive, or -equivocal tumor

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, as defined by 1 of the following:

  * Over 55 years of age with spontaneous cessation of menses for ≥ 1 year
  * 55 years of age and under with spontaneous cessation of menses for ≤ 1 year, but amenorrheic (e.g., spontaneous or secondary to hysterectomy) AND follicle-stimulating hormone level > 34.4 IU/L
  * Bilateral oophorectomy

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No recent unstable myocardial infarction
* No prior stroke
* No high blood pressure
* No other uncontrolled cardiovascular disease

Other

* Other prior malignancies without metastatic disease allowed
* Willing and able to complete quality of life questionnaires in either English or French
* No uncontrolled metabolic or endocrine disease
* No malabsorption syndrome

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 3 months since prior and no concurrent hormone replacement therapy or raloxifene
* At least 6 months since prior tamoxifen
* No concurrent steroid therapy
* No concurrent selective estrogen-receptor modulators
* No other concurrent endocrine or hormonal therapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2000-12-05 (Actual); Primary Completion 2007-11-16 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage change of the BMD parameters from baseline BMD values | 7 years
Percentage change of bone biomarker measurements (serum bone alkaline phosphatase and urine N-telopeptide) from baseline values | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (10):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
- Canada (8):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Hamilton Osteoporosis Diagnostic Services, Hamilton, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hotel Dieu de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cigler T, Tu D, Yaffe MJ, Findlay B, Verma S, Johnston D, Richardson H, Hu H, Qi S, Goss PE. A randomized, placebo-controlled trial (NCIC CTG MAP1) examining the effects of letrozole on mammographic breast density and other end organs in postmenopausal women. Breast Cancer Res Treat. 2010 Apr;120(2):427-35. doi: 10.1007/s10549-009-0662-0. Epub 2009 Dec 6. PMID 19967558